CLINICAL TRIAL: NCT05649644
Title: Sensorimotor Block Dynamics and Hemidiaphragmatic Palsy: A Randomized Superiority Trial Comparing Selective Trunk Block and Supraclavicular Brachial Plexus Block
Brief Title: Sensorimotor Block Dynamics and Hemidiaphragmatic Palsy: Selective Trunk Block vs Supraclavicular Brachial Plexus Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.219 SeTB vs SC BPB_RCT
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Sensorimotor Block Dynamics; Hemidiaphragmatic Palsy; Upper extremity surgery; Selective Trunk Block; Supraclavicular Brachial Plexus Block
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either USG SeTB or supraclavicular BPB. The randomization sequence will be generated using an online randomization software (www.randomization.com) and prepared by a third party (Research assistant) not involved with the study. The randomization sequence will be assigned as 1 = SeTB group and 2 = SCBPB group and the group allocation card will be sealed within an opaque envelop by a research assistant.
Who Masked: Participant, Outcomes Assessor
Masking Description: 1. Patients will be blinded to the group allocation. Patients will also be unable to view the ultrasound monitor during block placement.
  2. The research nurse (outcome assessor) will not be present in the procedure room during block placement and will be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective Trunk Block (SeTB) (Active Comparator): Patient who scheduled an upper extremity surgery involving anywhere from the proximal humerus to distal hand or surgery involving any combination of these regions and randomized in SeTB group will receive a SeTB.It will be performed through two skin punctures and as three separate injections to the three trunks of the brachial plexus.
  Interventions: Procedure: Selective Trunk Block (SeTB)
- Supraclavicular Brachial Plexus Block (SC BPB) (Active Comparator): Patient who scheduled an upper extremity surgery involving anywhere from the proximal humerus to distal hand or surgery involving any combination of these regions and randomized in SeTB group will receive a SC BPB. It will be performed using a single ultrasound window demonstrating the trunks and divisions of the brachial plexus in a superolateral position relative to the subclavian artery at the supraclavicular fossa.
  Interventions: Procedure: Supraclavicular Brachial Plexus Block (SC BPB)

INTERVENTIONS:
Procedure: Selective Trunk Block (SeTB) — Patient will lie supine on the examination couch with the ipsilateral arm in the neutral position (adducted), neck slightly extended and the head turned slightly to the contralateral side. After local anesthetic (LA) infiltration (1-2 ml lidocaine 1%), the nerve block needle will be inserted and placed within the interscalene groove. Then, a 7 ml of a 1:1 mixture of lidocaine 2% with 1:200,000 epinephrine and levobupivacaine 0.5% will be slowly injected in aliquots. After that, the tip will be redirected lateral to the middle trunk. A further 8 ml of the LA mixture will be injected after which the nerve block needle will be completely withdrawn. The transducer will then be manipulated to a sub-omohyoid position. After LA infiltration, the nerve block needle is inserted in-plane until the needle tip is positioned close to and lateral to (9-12 o'clock position) the inferior trunk. A 10 ml of the LA mixture is injected in small aliquots and the needle will be removed after the injection.
  Arms: Selective Trunk Block (SeTB)
Procedure: Supraclavicular Brachial Plexus Block (SC BPB) — Patient will lie supine on the examination couch with the ipsilateral arm in the neutral position (adducted), neck slightly extended and the head turned slightly to the contralateral side. Patient will receive a subcutaneous infiltration with 1-2 ml of 0.9% normal saline (NS) at the superior and middle trunk level after which the needle will be completely withdrawn. Then, a local anesthetic (LA) infiltration (1-2 ml lidocaine 1%) will then be performed at the supraclavicular fossa and the nerve block will be inserted in-plane to place the needle tip at the corner pocket. After that, 15-ml of a 1:1 mixture of lidocaine 2% with 1:200,000 epinephrine and levobupivacaine 0.5% will be slowly injected in aliquots. Once completed, the needle tip is gently withdrawn and redirected into the cluster formed by the divisions of brachial plexus. Then, the remaining 10-ml of the same LA mixture will be injected in small aliquots and the needle will be removed after the injection.
  Arms: Supraclavicular Brachial Plexus Block (SC BPB)

SUMMARY:
Ultrasound guided supraclavicular brachial plexus block (BPB) has been extensively studied and recommended as a sole anesthetic for upper extremity surgeries. The efficacy of ultrasound-guided (USG) SeTB for surgical anesthesia of the entire upper extremity and cadaver anatomic study evaluating the spread of the injectate after a simulated SeTB is further confirmed from the results of our previous research. Although the results in our previous study are encouraging, there is a paucity of data on sensorimotor blockade and incidence of hemidiaphragmatic palsy after a SeTB, and no data comparing SeTB with a supraclavicular BPB techniques which this study aims to evaluate. We hypothesise that USG SeTB is superior to supraclavicular BPB in anesthetising the entire upper extremity from the shoulder to hand.

DETAILED DESCRIPTION:
Ultrasound guided supraclavicular brachial plexus block (BPB) has been extensively studied and recommended as a sole anesthetic for upper extremity surgeries. The supraclavicular BPB is often touted to be the 'spinal of the upper extremity' as it produces anesthesia of the entire upper extremity except for the T2 dermatome.

However, based on clinical experience, such a claim is grossly unsubstantiated. This is evident from the finding that supraclavicular BPB is associated with 2-36% inferior trunk or ulnar nerve sparing. In addition, since the suprascapular nerve takes off more proximally from the superior trunk and the supraclavicular BPB is performed distally at the supraclavicular fossa, the effect of supraclavicular BPB on the suprascapular nerve, which predominantly supply the shoulder and proximal humerus, is not known and has not been objectively documented.

Nonetheless, supraclavicular BPB has been successfully used for shoulder surgery albeit with a large local anesthetic (LA) volume (50-60 ml) or combined with interscalene BPB, a hybrid BPB technique using 30-50 ml LA volume, for proximal humerus fracture surgeries. But such high LA volume is invariably associated with potential complications in the high risk population and therefore not used in contemporary clinical practice.

Since all major nerves supplying the upper extremity, including suprascapular nerve, passes through the trunks of the brachial plexus, we proposed that by selectively identifying and blocking the three trunks of the brachial plexus with small doses of LA-selective trunk block (SeTB), it is feasible to produce anesthesia of the entire upper extremity, i.e., from shoulder to hand. This is further confirmed from the results of our research evaluating the efficacy of ultrasound-guided (USG) SeTB for surgical anesthesia of the entire upper extremity and cadaver anatomic study evaluating the spread of the injectate after a simulated SeTB. Although these are encouraging results, there is a paucity of data on the sensorimotor blockade and incidence of hemidiaphragmatic palsy comparing SeTB and supraclavicular BPB techniques which this study aims to evaluate. We hypothesize that USG SeTB is superior to supraclavicular BPB in anesthetizing the entire upper extremity from shoulder to hand.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients
* Undergoing elective or emergency upper extremity surgery involving anywhere from the proximal humerus to distal hand or surgery involving any combination of these regions

Exclusion Criteria:

* Patient refusal
* Pregnancy
* Skin infection at the site of block placement
* History of allergy to local anaesthetic (LA) drugs
* Bleeding tendency or with evidence of coagulopathy
* Pre-existing respiratory disease
* Neurological deficit or neuromuscular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Readiness for surgery (Change of sensory and motor function from baseline to blockade) | Within 45 minutes after the block at 5 minutes interval
  When the patient is able to achieve a composite score of 20 out of 22 with a sensory blockade score of at least 9 out of 10.
  Sensory blockade:Loss of sensation to cold stimulus (ice cube) in the cutaneous distribution of the median, radial, ulnar, musculocutaneous and axillary nerves will be tested.Graded using a 3-points scale: 0 = able to feel touch and cold, 1= feel touch but not cold, 2 = feel neither touch nor cold.
  Motor blockade:The median, radial, ulnar, musculocutaneous, axillary and suprascapular nerves will be assessed.Graded using a 3-points scale: 0 = no block, 1 = paresis and 2 = paralysis.
Change of ipsilateral Hemidiaphragmatic (phrenic nerve) function from baseline to 30 minutes after SeTB | Before and 30 minutes after SeTB
  Reduction in diaphragmatic excursion of more than 75% of baseline, or no movement, or paradoxical movement will be considered as complete paresis. Reduction in diaphragmatic excursion of between 25% and 75% will be considered as partial paresis and diaphragmatic excursion of less than 25% will be considered as 'no paresis. Each test will be performed 3 times, and values will be averaged.

SECONDARY OUTCOMES:
Complete sensory block | Within 45 minutes after the block at 5 minutes interval
  Sensory blockade score of at least 9 out of 10. Loss of sensation to cold stimulus (ice cube) in the cutaneous distribution of the median, radial, ulnar, musculocutaneous and axillary nerves will be tested.
  Graded using a 3-points scale:
  0 = able to feel touch and cold, 1= feel touch but not cold, 2 = feel neither touch nor cold.
Motor blockade | Within 45 minutes after the block at 5 minutes interval
  Motor blockade of the suprascapular nerve, median, radial, ulnar, musculocutaneous, axillary and suprascapular nerves will be assessed.
  Graded using a 3-points scale:
  0 = no block, 1 = paresis and 2 = paralysis.
Any occurrence of paradoxical movement | Within 45 minutes after the block
  Any paradoxical movement after the block will be documented.
Block performance time | Within 30 minutes after entering the procedure room
  The time taken from the start of the local anaesthetic (LA) skin infiltration to the end of the LA injection for the block.
Any occurrence of paresthesia | Immediately after the end of the block
  Any paresthesia experienced during the block will be assessed and recorded as a 'yes' or 'no' response.
Discomfort score | Immediately after the end of the block]
  Discomfort experienced during the regional anesthesia using a numeric rating scale (NRS, 0 to 100, 0=no discomfort, 100=extreme discomfort)
Any occurrence of symptomatic dyspnea | During and within 45 minutes after the block
  Any dyspnea experienced during and after the block will be assessed and recorded as a 'yes' or 'no' response.
Name and dosage of used rescue analgesia | During surgery
  Any rescue intravenous analgesic requirements during surgery will be documented with name and dosage.
Total amount of local anesthetic infiltration used | During surgery
  Any rescue LA infiltration requirements during surgery will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, New Territories,, Hong Kong, Hong Kong